CLINICAL TRIAL: NCT06770673
Title: Culturally Grounded Diabetes Intervention With Lakota Populations in South Dakota
Brief Title: Together Overcoming Diabetes - Great Plains
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: The NIH Community Engagement Alliance (Unknown); Oyate Health Center (Unknown); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00029399; OT2HL158287 (NIH)
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Waitlist randomized control trial
Who Masked: Outcomes Assessor
Masking Description: Independent Evaluators are masked to the study participants' randomized group status/
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Together Overcoming Diabetes Intervention (Experimental): Together Overcoming Diabetes curriculum adapted for Lakota caregivers and the caregivers families
  Interventions: Behavioral: TOD Great Plains
- Waitlist Standard of Care (Placebo Comparator): Participants who are waitlisted to receive the TOD intervention will receive Standard of Care.
  Interventions: Behavioral: Waitlist Standard of Care

INTERVENTIONS:
Behavioral: TOD Great Plains — The adapted TOD intervention is rooted in the original TOD structure, delivery system, and home-visiting teaching schedule. Local enhancements include intervention topics and activities to address local adult caregivers' diabetes management and to promote families' modifiable risk and protective factors targeted by this proposal and informed by the Wicozani wellness concept and measurement. The TOD intervention includes targeted content taught approximately bi-weekly by family health coaches over a 16-week period.
  Arms: Together Overcoming Diabetes Intervention
Behavioral: Waitlist Standard of Care — Participants who are waitlisted to receive the TOD intervention will receive Standard of Care.
  Arms: Waitlist Standard of Care

SUMMARY:
The goal of this research is to evaluate a scientifically rigorous diabetes intervention, Together Overcoming Diabetes (TOD), that has been tailored to address the unique underlying risk and protective factors and social determinants of diabetes among American Indian/Alaska Native (AI/AN) populations.

ELIGIBILITY:
Inclusion Criteria - Adult Index Participants:

* 18 years and older
* Self-identifies as American Indian or Alaska Native
* Rapid City-based participants who reside within 1 hour transportation range of the Oyate Health Center
* Verification from a health provider to confirm Type 2 Diabetes diagnosis by laboratory test.
* Caregiver to a 10- to 25-year-old in their home at the time of screening.
* Willing to complete all implementation and follow-up assessments.
* Willing to be randomized for the intervention.

Exclusion Criteria - Adult Index Participants:

* Inability to participate in full intervention or evaluation (e.g., planned move, residential treatment, etc.)
* Willing to serve as 'support person' for the adult participant.
* Has a circumstance that might impact successful participation based on provider judgment considering instances where diabetes control can become more difficult with advanced disease or special conditions including: pregnant, nursing, or planning to become pregnant, end-stage renal disease on dialysis, diabetes due to secondary causes such as Cushing's or Cystic Fibrosis, or any condition that may inhibit participation

Inclusion Criteria - Youth Support Participants:

* Between 10 years and 25 years old
* Self-identifies as American Indian or Alaska Native.
* Willing to serve as 'support person' for the adult participant.
* Willing to complete all implementation and follow-up assessments.
* Willing to be randomized for the intervention.

Exclusion Criteria - Youth Support Participants:

* Cognitively or visually impaired
* Youth in foster care (due to potential mobility of foster youth).

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Glycated hemoglobin (HbA1c) | Baseline, 3 months, 6 months, and 12 months
  Glycated hemoglobin as measured by a point-of-care A1c test

CONTACTS AND LOCATIONS:
Overall Officials: Donald Warne, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Center for Indigenous Health - Great Plains Hub, Rapid City, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No